CLINICAL TRIAL: NCT03722225
Title: Carbohydrate Loading Before and Intermittent High Carbohydrate Intake During Prolonged Physical Exercise in Individuals With Type 1 Diabetes is Associated With Good Glucose Control
Brief Title: CHO-loading Before and High Intermittent CHO-intake During Physical Exercise in T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Dnr:2012/159
Record Dates: First submitted 2018-10-18; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate Loading

STUDY DESIGN:
Intervention Model Description: This is a descriptive, single arm, non-randomized interventional study. The intervention consisted of carbohydrate loading prior to and intermittent high carbohydrate intake during physical exercise and a proactive use of Real-Time Continuous Glucose Monitoring (rtCGM) to achieve and maintain glucose control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Descriptive, single arm, interventional study (Experimental): The intervention consisted of carbohydrate loading prior to and intermittent high carbohydrate intake during physical exercise and a proactive use of Real-Time Continuous Glucose Monitoring (rtCGM) to achieve and maintain glucose control
  Interventions: Other: Carbohydrate loading and high intermittent carbohydrate intake during physical exercise

INTERVENTIONS:
Other: Carbohydrate loading and high intermittent carbohydrate intake during physical exercise — The intervention consisted of carbohydrate loading prior to and intermittent high carbohydrate intake during PE and a proactive use of Real-Time Continuous Glucose Monitoring (rtCGM) to achieve and maintain glucose control

SUMMARY:
Prolonged physical exercise (PE) is a challenge in type 1 diabetes with an increased incidence of both hypoglycemia and hyperglycemia.

The purpose was to evaluate the impact of two consecutive days of carbohydrate (CHO) loading, followed by high intermittent CHO-intake during prolonged PE, facilitated by a proactive use of Real-Time Continuous Glucose Monitoring (rtCGM), on glucose control in individuals with type 1 diabetes.

Ten physically active individuals with type 1 diabetes were invited to participate in a 3-day long sports camp with the objective to evaluate CHO-loading and high intermittent CHO-intake during prolonged PE. 1.5 months later the same procedure was evaluated during a 90 km cross-country skiing race. Participants were instructed to act proactively using rtCGM with predictive alerts set for high and low glucose values to maintain sensor glucose values within target range, defined as 72-180 mg/dl (4-10 mmol/l).

DETAILED DESCRIPTION:
This is a descriptive, single arm, non-randomized interventional study. The intervention consisted of carbohydrate loading prior to and intermittent high carbohydrate intake during physical exercise and a proactive use of Real-Time Continuous Glucose Monitoring (rtCGM) to achieve and maintain glucose control.

Central Contact Person Stig A Mattsson, dietician PhD student Phone: +46702047759 E-mail: stigmattsson@live.com

IPD Sharing Statement No: There is not a plan to make IPD available.

ELIGIBILITY:
Inclusion criteria:

* age 18-50 years
* type 1 diabetes
* diabetes duration >1 year
* exercising regularly ≥3 workout/week
* previous experience from cross-country skiing

Exclusion Criteria:

* A1c 8.6% NGSP (70 mmol/mol IFCC)
* proliferative retinopathy
* known nephropathy
* cardiac failure
* following a low-carbohydrate diet.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-25 (Actual)

PRIMARY OUTCOMES:
The percentage of the glucose values spent in target range, defined as 72-180 mg/dl. | Through 48 hours of carbohydrate loading and an average of 6.5 hours of cross-country skiing.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Jendle, professor, Principal Investigator — Institute of Medical Sciences, Örebro University, 701 82, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
We will not share participants' data with other researchers.

REFERENCES:
- [Derived] Mattsson S, Jendle J, Adolfsson P. Carbohydrate Loading Followed by High Carbohydrate Intake During Prolonged Physical Exercise and Its Impact on Glucose Control in Individuals With Diabetes Type 1-An Exploratory Study. Front Endocrinol (Lausanne). 2019 Aug 21;10:571. doi: 10.3389/fendo.2019.00571. eCollection 2019. PMID 31496994